CLINICAL TRIAL: NCT04958863
Title: Running and Facemasks During COVID-19 Pandemic: a Randomized Crossover Trial
Brief Title: Impact of Facemasks on Running During COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Juan Pablo Martinez, Orthopaedic surgeon, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1718
Record Dates: First submitted 2021-06-30; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Shortness of Breath
Keywords: Oxymetry; Shortness of Breath; Running; Masks; COVID-19
MeSH Terms: conditions — Dyspnea; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Mask (No Intervention): Runners do not use mask while running
- Surgical Mask (Experimental): Runners use surgical mask while running
  Interventions: Other: Surgical mask
- Polyester Reusable Mask (Experimental): Runners use polyester reusable mask while running
  Interventions: Other: Polyester reusable mask

INTERVENTIONS:
Other: Surgical mask — Use of a surgical mask during test
  Arms: Surgical Mask
Other: Polyester reusable mask — Use of a polyester reusable mask during test
  Arms: Polyester Reusable Mask

SUMMARY:
Randomized crossover clinical trial in which a group of runners are ask to complete a 15 minutes standardized physical test on a treadmill. The same group of participants are randomized to the order in which they use a facemask (surgical mask, polyester reusable cloth mask) or no mask, while running.

Each test, according to the type of mask or no mask, are held on different dates. Heart rate, oxygen saturation and shortness of breath are measured every 3 minutes during the test.

DETAILED DESCRIPTION:
Between 15-20 recreational runners are included in a crossover trial to run under three different conditions the same 15-minutes treadmill running test. They Will run wtih surgical mask, polyester reusable cloth mask or without mask. The order in which they use or not the mask is randomized. Each test is done on a different day.

Heart rate, oxygen saturation and shortness of breath are measured every 3 minutes during the test.

The primary outcomes are the differences in heart rate, oxygen saturation and shortness of breath at the end of the test, between groups.

ELIGIBILITY:
Inclusion Criteria:

* Recreational runners.
* Age between 16-65 years.
* Workers or students from the health area.

Exclusion Criteria:

* None.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Shortness of breath in a visual analogue score (1-10) | At the end of the 15-minutes test
  The difference in the subjective sensation of shortness of breath between groups at the end of the test
Oxygen saturation | At the end of the 15-minutes test
  The difference in the measured oxygen saturation with pulse oxymetry between groups at the end of the test
Heart rate | At the end of the 15-minutes test
  The difference in the measured heart rate with pulse oxymetry between groups at the end of the test

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Martinez, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No